CLINICAL TRIAL: NCT00117195
Title: Open-Label Validation Study of Neurophysiologic Changes in Individuals With Parkinson's Disease, at Risk for Parkinson's Disease and Healthy Controls
Brief Title: A Study of Neurophysiologic Changes in Individuals With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Molecular NeuroImaging (Other)
Responsible Party: Principal Investigator, Kenneth Marek, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Other Study IDs: Neurophysiologic; Neurophys (Other: MNI/IND)
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Parkinson's Disease; Parkinsonian Syndrome
Keywords: parkinson; diagnosis; screening
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In addition, the study will evaluate serum samples for changes in proteins or metabolites that may be indicators of early changes associated with Parkinson's disease or parkinsonian syndrome.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PD/PS
  Interventions: Device: Automated Neuropsychological Assessment Matrix

INTERVENTIONS:
Device: Automated Neuropsychological Assessment Matrix — This study will evaluate a profile of neurophysiologic tests for potentially predictive signs of PD or PS in individuals with PD or PS, those who may be at risk for PD or PS and in a population of individuals without parkinsonian symptoms or any other neurologic conditions.
  In addition, the study will evaluate serum samples for changes in proteins or metabolites that may be indicators of early changes associated with Parkinson's disease or parkinsonian syndrome.

SUMMARY:
The goal of this study is to investigate neurophysiologic tests that have the potential of serving as screening tools for Parkinson's disease. These neurophysiologic tests will be administered to individuals with Parkinson's disease and parkinsonian syndrome and validated against a healthy control population.

Specifically, this study will look at changes in motor function, cognitive function, handwriting, speech, and olfactory function in individuals with Parkinson's disease, individuals at risk for Parkinson's disease and healthy controls.

DETAILED DESCRIPTION:
One of the greatest challenges in Parkinson's research is the identification of individuals who are at risk or have early Parkinson's disease (PD) or parkinsonian syndrome (PS). Subtle signs that do not meet the diagnostic criteria for PD may occur during this period.

This study will evaluate a profile of neurophysiologic tests for potentially predictive signs of PD or PS in individuals with PD or PS, those who may be at risk for PD or PS and in a population of individuals without parkinsonian symptoms or any other neurologic conditions.

In addition, the study will evaluate serum samples for changes in proteins or metabolites that may be indicators of early changes associated with Parkinson's disease or parkinsonian syndrome.

Each study participant will be scheduled for a 90 minute study visit.

This visit may include the following procedures:

* Screening for eligibility
* Clinical assessments
* Neurological evaluation
* Computerized cognitive testing
* Olfactory testing
* Computerized handwriting testing
* Speech evaluation
* Blood sample for biochemical and/or genetic analysis

The study will be conducted at the Institute for Neurodegenerative Disorders (IND), which is a not for profit research institute specializing in Parkinson's disease research.

Clinical data will be collected, stored and analyzed at IND to evaluate whether there are significant differences between the performance of the parkinsonian study participants, individuals with risk factors for PD or PS, and the healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

As a participant with PD or PS:

* Age >21
* Clinical diagnosis of PD or PS (at least two of the three cardinal symptoms: resting tremor, rigidity, bradykinesia) and a clinical response to dopaminergic therapy

For Healthy Control:

* Age >21

Exclusion Criteria:

As a participant with PD or PS:

* Any other concomitant neurologic condition likely to interfere with handwriting, use of the computer, or other motor tasks tested in this study (e.g. stroke, demyelinating disease, visual loss)

For Healthy Control:

* Any indication of parkinsonism on examination
* Any other concomitant neurologic condition likely to interfere with handwriting, use of the computer, or other motor tasks (e.g. stroke, demyelinating disease, visual loss)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: These neurophysiologic tests will be administered to individuals with Parkinson's disease and parkinsonian syndrome and validated against a healthy control population.
Sampling Method: Non-Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2003-05; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Marek, MD, Principal Investigator — Institute for Neurodegenerative Disorders; Laura Leary, Study Director — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- [Background] Agid Y, Javoy-Agid, Ruberg M. Biochemistry of neurotransmitters in Parkinson's disease. In: Marsden CD, Fahn S, eds. Movement Disorders 2: neurology, vol 7. London: Butterworths, pp 166-230.
- [Background] Blandini F, Mangiagalli A, Cosentino M, Marino F, Samuele A, Rasini E, Fancellu R, Martignoni E, Riboldazzi G, Calandrella D, Frigo GM, Nappi G. Peripheral markers of apoptosis in Parkinson's disease: the effect of dopaminergic drugs. Ann N Y Acad Sci. 2003 Dec;1010:675-8. doi: 10.1196/annals.1299.123. PMID 15033810
- [Background] Bleiberg J, Kane RL, Reeves DL, Garmoe WS, Halpern E. Factor analysis of computerized and traditional tests used in mild brain injury research. Clin Neuropsychol. 2000 Aug;14(3):287-94. doi: 10.1076/1385-4046(200008)14:3;1-P;FT287. PMID 11262703
- [Background] Brin MF, Fahn S, Blitzer A, Ramig LO, Stewart CF. (1992) Movement disorders of the larynx. In: Blitzer AA, Brin MF, Fahn S, Sasaki CT Harris K eds. Neurological disorders of the larynx. New York: Thieme Medical, pp 248-78.
- [Background] Critchley EM. Speech disorders of Parkinsonism: a review. J Neurol Neurosurg Psychiatry. 1981 Sep;44(9):751-8. doi: 10.1136/jnnp.44.9.751. PMID 7031185
- [Background] Darley FL, Aronson AE, Brown JR. Clusters of deviant speech dimensions in the dysarthrias. J Speech Hear Res. 1969 Sep;12(3):462-96. doi: 10.1044/jshr.1203.462. No abstract available. PMID 5811846
- [Background] Fahn S. (1986) Parkinson's disease and other basal ganglia disorders. In Asbiry AK, Mchann GM, McDonald WI, eds. Diseases of the nervous system: clinical neurobiology. Philadelphia: Ardmore Medical Books, pp1217-1228.
- [Background] Koller WC, Montgomery EB. Issues in the early diagnosis of Parkinson's disease. Neurology. 1997 Jul;49(1 Suppl 1):S10-25. doi: 10.1212/wnl.49.1_suppl_1.s10. PMID 9222271
- [Background] Lees AJ, Smith E. Cognitive deficits in the early stages of Parkinson's disease. Brain. 1983 Jun;106 (Pt 2):257-70. doi: 10.1093/brain/106.2.257. PMID 6850270
- [Background] Levin BE, Llabre MM, Weiner WJ. Cognitive impairments associated with early Parkinson's disease. Neurology. 1989 Apr;39(4):557-61. doi: 10.1212/wnl.39.4.557. PMID 2927680
- [Background] Logemann JA, Fisher HB, Boshes B, Blonsky ER. Frequency and cooccurrence of vocal tract dysfunctions in the speech of a large sample of Parkinson patients. J Speech Hear Disord. 1978 Feb;43(1):47-57. doi: 10.1044/jshd.4301.47. PMID 633872
- [Background] Pillon B, Ertle S, Deweer B, Bonnet AM, Vidailhet M, Dubois B. Memory for spatial location in 'de novo' parkinsonian patients. Neuropsychologia. 1997 Mar;35(3):221-8. doi: 10.1016/s0028-3932(96)00091-7. PMID 9051671
- [Background] Pirozzolo FJ, Hansch EC, Mortimer JA, Webster DD, Kuskowski MA. Dementia in Parkinson disease: a neuropsychological analysis. Brain Cogn. 1982 Jan;1(1):71-83. doi: 10.1016/0278-2626(82)90007-0. PMID 6927555
- [Background] Polymeropoulos MH, Lavedan C, Leroy E, Ide SE, Dehejia A, Dutra A, Pike B, Root H, Rubenstein J, Boyer R, Stenroos ES, Chandrasekharappa S, Athanassiadou A, Papapetropoulos T, Johnson WG, Lazzarini AM, Duvoisin RC, Di Iorio G, Golbe LI, Nussbaum RL. Mutation in the alpha-synuclein gene identified in families with Parkinson's disease. Science. 1997 Jun 27;276(5321):2045-7. doi: 10.1126/science.276.5321.2045. PMID 9197268
- [Background] Ramig LO. (1993) Speech therapy for patients with Parkinson's disease. NCVS Status Prog Rep 5:83-90.
- [Background] Tetrud JW. Preclinical Parkinson's disease: detection of motor and nonmotor manifestations. Neurology. 1991 May;41(5 Suppl 2):69-71; discussion 72. doi: 10.1212/wnl.41.5_suppl_2.69. PMID 2041596